CLINICAL TRIAL: NCT04086264
Title: A Phase 1b/2 Study of IMGN632 as Monotherapy or Combination With Venetoclax and/or Azacitidine for Participants With CD123-Positive Acute Myeloid Leukemia
Brief Title: IMGN632 as Monotherapy or With Venetoclax and/or Azacitidine for Participants With CD123-Positive Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMGN632-0802; 2024-514197-50-00 (Other: EU CT)
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; AML; Minimal detectable disease; MRD; CD123; Relapsed/refractory; Frontline
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Azacitidine; Decitabine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Regimen A (Closed to Enrollment) (Experimental): IMGN632, administered intravenously on Day 7 of a 28 day cycle at 0.015 mg/kg, 0.045 mg/kg, or 0.09 mg/kg, in combination with azacitidine, administered subcutaneously or intravenously daily at 75 mg/m2 on Days 1 to 7 of a 28 day cycle. Cycle 1 azacitidine dose in subsequent cohorts may be reduced.
  Interventions: Drug: Azacitidine; Drug: IMGN632
- Regimen B (Closed to Enrollment) (Experimental): IMGN632, administered intravenously on Day 7 of a 21 day cycle at 0.015 mg/kg, 0.045 mg/kg, or 0.09 mg/kg, in combination with venetoclax, administered orally daily at 100 mg on Day 1, 200mg on Day 2, and 400 mg on the day 3 up to Day 21 of a 21 day cycle. Alternate schedules with reduced venetoclax administration may be explored.
  Interventions: Drug: IMGN632; Drug: Venetoclax
- Regimen C-Frontline&Relapsed/Refractory(Closed to Enrollment) (Experimental): IMGN632, administered intravenously on Day 7 of a 28 day cycle at 0.015 mg/kg or 0.045 mg/ kg, in combination with azacitidine, administered subcutaneously or intravenously daily at 35-75 mg/ m2 given for Days 1 to 7 of a 28 day cycle and venetoclax, administered orally daily at 100 mg on Day 1, 200mg on Day 2, and 400 mg on Day 3 up to Day 28 of a 28 day cycle. Alternate schedules with reduced venetoclax administration or reduced azacitidine dose or administration may be explored.
  Interventions: Drug: Azacitidine; Drug: IMGN632; Drug: Venetoclax
- Regimen D (Closed to Enrollment) (Experimental): IMGN632, administered intravenously on Day 1 of a 21 day cycle at 0.045 mg/kg, as a monotherapy for Fit and Unfit MRD+ patients.
  Interventions: Drug: IMGN632

INTERVENTIONS:
Drug: Azacitidine — Commercially available formulation given subcutaneously (SC) or intravenous (IV)
  Other Names: Vidaza; Decitabine
  Arms: Regimen A (Closed to Enrollment); Regimen C-Frontline&Relapsed/Refractory(Closed to Enrollment)
Drug: IMGN632 — Study formulation given intravenously (IV)
  Other Names: CD123-targeted ADC
Drug: Venetoclax — Commercially available formulation administered orally
  Other Names: Venclexta; Venclyxto
  Arms: Regimen B (Closed to Enrollment); Regimen C-Frontline&Relapsed/Refractory(Closed to Enrollment)

SUMMARY:
This is an open-label, multicenter, Phase 1b/2 study to determine the safety and tolerability of IMGN632 and assess the antileukemia activity of IMGN632 when administered in combination with azacitidine and/or venetoclax in participants with relapsed and frontline CD123-positive AML.

DETAILED DESCRIPTION:
This study explores multiple IMGN632 doses in combination and monotherapy Regimens, including (A - closed to enrollment)) azacitidine, (B-closed to enrollment) venetoclax, (C) azacitidine+venetoclax, and (D- closed to enrollment) monotherapy in MRD+ AML. For combination Regimens A-C, a Phase 1b Dose Escalation Cohort will determine the recommended Phase 2 dose (RP2D) of IMGN632 in that specific combination Regimen, followed by a Phase 2 Dose Expansion Cohort for each combination Regimen to characterize the safety profile further and assess the antileukemia activity of the different combination Regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 18 years of age.
* Patients must have confirmed diagnosis of AML (excluding acute promyelocytic leukemia) based on World Health Organization classification (Arber 2016).
* Disease characteristics and allowable prior therapy:

  * Patients must be evaluated for any available standard of care therapies (including induction, consolidation chemotherapy and/or transplant) and, in the opinion of the treating physician, be deemed appropriate for this experimental therapy.
  * Treatment-naïve (untreated) patients will be allowed in the Expansion Phase for Regimen C (Triplet) (IMGN632 + azacitidine + venetoclax). No prior treatments with hypomethylating agents (HMAs) for MDS are allowed.
  * Patients must have CD123-positive AML as confirmed by local flow cytometry (or immunohistochemistry [IHC]).
  * Patients may have received prior CD123-targeted therapies, except IMGN632, as long as CD123 remains detectable during screening.
  * Relapsed or refractory CD123-positive AML patients will be allowed to enroll in the Escalation Phase of Regimens A, B, and C (Triplet (IMGN632 + azacitidine, venetoclax, or azacitidine + venetoclax, respectively) and relapsed CD123-positive AML patients will be allowed to enroll the Expansion Phase of Regimens A-C. Note: Patients may also have received up to 2 prior lines of therapy, eg, frontline treatment (induction, consolidation [including transplant], and maintenance) and 1 salvage regimen.
  * Patients enrolling in Regimen D must be in CR (CR/CRh/CRp/ CRi) and be MRD+ at the time of screening, confirmed by central laboratory testing. Patients may have no more than 2 prior lines of therapy (which may include stem cell transplant), ie, frontline or first salvage. Note: Fit patients who received intensive treatment (eg 3+7, HiDAC) are eligible for Regimen D Cohort D1. Unfit patients who received non-intensive treatment (eg, HMA, low dose cytarabine) are eligible for Regimen D Cohort D2.
* Previous treatment-related toxicities must have resolved to Grade 1 or baseline (excluding alopecia).
* For patients enrolling in Regimens A-D, total WBC count must < 25 × 10^9 cells/L. Hydroxyurea may be used to control blood counts before Cycle 1 Day 1, at the discretion of the treating physician, according to institutional practice. During the Escalation Phase in Regimens A-C, hydroxyurea may also be used during Cycle 1.
* Liver enzymes (AST and ALT) ≤ 3 × the upper limit of normal (ULN).
* Total bilirubin ≤ 1.5 × the ULN; patients with Gilbert syndrome must have total bilirubin < 3.0 × ULN with direct bilirubin < 1.0 × ULN at the time of enrollment.
* An estimated glomerular filtration rate (eGFR) of > 30 mL/min/1.73 m2 or creatinine clearance of > 30 mL/min.
* Left ventricular ejection fraction (LVEF) ≥ 45% for patients enrolling in Regimens A-D based on locally available assessment, eg, echocardiogram or other modality.
* Patients with prior autologous or allogeneic bone marrow transplant are eligible. Patients with an allogeneic transplant must meet the following conditions: The transplant must have been performed more than 120 days before the date of dosing on this study, the patient must not have active ≥ Grade 2 graft versus host disease (GvHD), or extensive chronic GvHD of any severity, and must be off all immunosuppression for at least 2 weeks prior to first dose of IMGN632.
* Participants or their legally authorized representative must voluntarily sign and date an informed consent, approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC), before performance of any study-related procedure not part of normal medical care.
* Women of childbearing potential (WCBP), defined as sexually mature women who have not undergone surgical sterilization or who have not been naturally postmenopausal for at least 12 consecutive months (ie, who have had menses any time in the preceding 12 consecutive months), must agree to use acceptable contraceptive methods while on study drug and for at least 7 months after the last dose of IMGN632.
* WCBP must have a negative pregnancy test within 3 days before the first dose of study drug.
* Male patients who are able to father children must agree to use acceptable methods of contraception throughout the study and for at least 4 months after the last dose of study drug(s).
* Patients with prior malignancy are eligible; however, the patient's malignancy must be well-controlled or stable and have completed all systemic chemotherapy and radiotherapy for the prior malignancy at least 6 months before enrollment, and all treatment-related toxicities must have resolved to ≤ Grade 1 (excluding alopecia). Note: patients with prostate cancer or breast cancer on adjuvant hormonal therapy are eligible and may or may not be on long-term maintenance treatment that is unlikely to interfere with study therapy. Note: patients with tumors with a negligible risk for metastasis or death (eg, adequately controlled basal cell carcinoma or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast) are eligible.
* Patients in expansion Cohorts C1 and C2 must be considered ineligible for intensive induction therapy defined by the following:

  * ≥ 75 years of age OR
  * < 75 years of age with at least one of the following co-morbidities documented within 28 days of Cycle 1 Day 1:
  * ECOG performance status of 2 or 3
  * History of congestive heart failure requirement treatment or ejection fraction ≤ 50% or chronic stable angina
  * Diffusing capacity of the lung for carbon monoxide ≤ 65% or forced expiratory volume in 1 second ≤ 65%
  * Creatinine clearance ≥ 30 mL/min to < 45 mL/min
  * Moderate hepatic impairment with total bilirubin > 1.5 to ≤ 3.0 × ULN
* Patients in Cohort C1 and C2 must have an ECOG performance status of 0 to 2 for those ≥ 75 years of age OR 0 to 3 for < 75 years of age.
* Patients must not be incarcerated and must be freely willing and able to provide informed consent. Examples of patients unable to freely provide informed consent may include some adults under legal protection measure (eg, under guardianship/curatorship) or unable to express their consent and select adults under psychiatric care. Investigator's discretion should be applied.

Exclusion Criteria:

* Patients who have received any anticancer therapy, including investigational agents, within 14 days (or within 28 days for checkpoint inhibitors) before drug administration on this study (hydroxyurea is allowed before beginning study treatment). Patients must have recovered to baseline from all acute toxicity from this prior therapy.
* Patients who have been previously treated with IMGN632.
* Patients with myeloproliferative neoplasm-related secondary AML are excluded from the Dose Expansion Phase of the study.
* Patients with active central nervous system (CNS) AML will be excluded. A lumbar puncture does not need to be performed unless there is clinical suspicion of CNS involvement per investigator judgement. Concurrent therapy for CNS prophylaxis or continuation of therapy for controlled CNS AML is allowed with the approval of the sponsor.
* Patients with a history of sinusoidal obstruction syndrome/venous occlusive disease of the liver.
* Myocardial infarction within 6 months before enrollment or New York Heart Association Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities before study entry.
* Clinically relevant active infection including known active hepatitis B or C, HIV infection, or cytomegalovirus or any other known concurrent infectious disease that, in the judgment of the investigator, would make a patient inappropriate for enrollment into this study (testing not required).
* Patients who have undergone a major surgery within 4 weeks (or longer if not fully recovered) before study enrollment.
* Serious or poorly controlled medical conditions that could be exacerbated by treatment or that would seriously compromise safety assessment or compliance with the protocol, in the judgment of the investigator.
* Women who are pregnant or breastfeeding
* Prior known hypersensitivity reactions to monoclonal antibodies (≥ Grade 3).
* Prior known hypersensitivity reactions to study drugs and/or any of their excipients.
* Patients who have a history of allergy to IMGN632 (or any of its excipients), azacitidine, or venetoclax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | approximately 3 years
  Evaluate the safety and tolerability and identify an RP2D of IMGN632 when administered in combination with azacitidine, with venetoclax, and with azacitidine and venetoclax in patients with relapsed or refractory CD123-positive AML through review of Treatment Emergent Adverse Events and abnormal laboratory values that result in a failure to meet the criteria for re-treatment.
Preliminary antileukemia activity | approximately 20 months
  Assess preliminary antileukemia activity of IMGN632 when administered as a monotherapy in MRD+ Fit and MRD + Unfit AML patient populations, and in combination with azacitidine, with venetoclax, and with azacitidine and venetoclax in patients with relapsed or untreated AML as assessed by complete response, complete remission with partial hematologic recovery, complete remission with incomplete platelet recovery, morphologic leukemia-free state, partial response, and duration of remission.
Minimal Residual Disease Levels | approximately 18 months
  Assess Minimal Residual Disease Levels using central flow cytometry-based testing.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) (Dose Expansion Phase) | Up to approximately 12 months
Study Drug Concentration (Dose Escalation and Expansion) | Up to approximately 12 months
Anti-drug Antibody Concentration (Dose Escalation and Expansion) | Up to approximately 12 months
Minimal Residual Disease Levels (Dose Escalation) | Up to approximately 7 months

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (29):
- United States (13):
  - City of Hope National Medical Center /ID# 269273, Duarte, California
  - University Of California Irvine Medical Center /ID# 269275, Orange, California
  - Moffitt Cancer Center /ID# 269269, Tampa, Florida
  - Northwestern University- Robert H. Lurie Comprehensive Cancer Center /ID# 269642, Chicago, Illinois
  - Dana-Farber Cancer Institute /ID# 269267, Boston, Massachusetts
  - University of Michigan /ID# 269079, Ann Arbor, Michigan
  - Mayo Clinic Hospital Rochester /ID# 269643, Rochester, Minnesota
  - Roswell Park Cancer Institute /ID# 269266, Buffalo, New York
  - New York Presbyterian Hospital Weill Cornell Medical Center /ID# 269271, New York, New York
  - Duke University Health System /ID# 269268, Durham, North Carolina
  - Cleveland Clinic - Cleveland /ID# 269272, Cleveland, Ohio
  - MD Anderson Houston /ID# 269265, Houston, Texas
  - Fred Hutchinson Cancer Research Center /ID# 269270, Seattle, Washington
- France (6):
  - Institut Paoli-Calmettes /ID# 269080, Marseille, Bouches-du-Rhone
  - IUCT Oncopole /ID# 269284, Toulouse, Occitanie
  - Hôpital Saint-Louis /ID# 269282, Paris, Paris
  - Centre Antoine-Lacassagne /ID# 269285, Nice, Provence-Alpes-Côte d'Azur Region
  - Hospices Civils de Lyon - Centre Hospitalier Lyon-Sud /ID# 269286, Pierre-Bénite, Rhone
  - Centre Hospitalier de Versailles André Mignot /ID# 269287, Le Chesnay
- Germany (3):
  - Universitaetsklinikum Ulm /ID# 269686, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Muenster /ID# 269688, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig /ID# 269682, Leipzig, Saxony
- Italy (4):
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 269281, Bologna, Bologna
  - Istituto Europeo Di Oncologia /ID# 269646, Milan, Milano
  - Azienda Ospedaliero Universitaria Maggiore Della Carità /ID# 269280, Novara, Novara
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST - IRCCS /ID# 269279, Meldola, Reggio Emilia
- Spain (2):
  - Hospital MD Anderson Cancer Center Madrid /ID# 269641, Madrid, Madrid
  - Hospital Universitario y Politecnico La Fe /ID# 269278, Valencia, Valencia
- Oxford University Hospital NHS Trust /ID# 269647, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=IMGN632-0802